CLINICAL TRIAL: NCT03584061
Title: Treatment of Chronic Postherpetic Pain With Fat Grafting - A Pilot Study
Brief Title: Treatment of Chronic Postherpetic Pain With Fat Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sollie, Principal investigator, M.D, Dept. of Plastic and Reconstructive Surgery, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20180007
Record Dates: First submitted 2018-05-01; First posted 2018-07-12 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Post Herpetic Neuralgia; Herpes Zoster
Keywords: Chronic Pain; Herpes Zoster; Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: The five patients included will all receive a fat graft in the area affected by PHN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fat grafting/fat transplant. (Experimental): Each patient receives fat grafting to the site of dermal pain. Fat is to be harvested for either the abdomen or the thigh.
  Interventions: Procedure: Fat grafting

INTERVENTIONS:
Procedure: Fat grafting — The area of dermal pain is identified and marked prior to surgery. The surgery starts with liposuction, either on the abdomen or the thigh. The harvested fat is prepared for fat grafting by sedimenting it for 10 minutes. The fat is then injected into the painful area, marked pre-surgery.
  Other Names: Fat transplant, lipofilling

SUMMARY:
This study evaluates the possible beneficial effect of fat grafting for post herpetic neuralgia.

DETAILED DESCRIPTION:
Herpes Zoster (HZ),is a condition caused by Varizella-Zooster virus (VZV), The disease is caused by reactivation of a latent VZV-infection in the sensory ganglia.

Clinically the condition is characterized by a painful, unilateral, vesicular rash. Pain is the most prominent symptom in around 90% of patients. In 10% of patients this pain remains and becomes chronic.

Post-herpetic neuralgia is a chronic pain syndrome that occurs after the dermal manifestations disappears.

Treatment is complex and mainly topical or systemic. For many patients this is not sufficient and they live with constant pain.

Fat grafting has shown promise in treating several different painful conditions such as post mastectomy pain syndrome, painful scars etc.

This study investigates is PHN can be treated by fat grafting.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Pain in area of former VZV-infection.
* Pain present over 3 months after reactivation of VZV and is present at least 4 days a week and of intensity >3 on the VAS-scale.

Exclusion Criteria:

* Psychiatric illness that could potentially affect the study.
* Other indication for fat grafting than pain.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain [LEVEL OF PAIN] | 6 months
  Neuropathic Pain Symptom inventory (NPSI), Questionnaire. NPSI consists of 12 items in total: 10 items investigates differential symptoms descriptors and 2 items evaluate spontaneous and paroxysmal spontaneous pain.
  The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of the 10 descriptors.
  The descriptors are:
  Burning, Squeezing, Pressure, Electric Shocks, Stabbing, Provoked by brushing. Provoked by pressure, Evoked by cold stimulation, Pins and needles, Tingling.

SECONDARY OUTCOMES:
Quality of life [QUALITY OF LIFE/ SATISFACTION] | 6 months
  Short Form 36 (SF-36), Questionnaire. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per a scoring key. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. After this, items in the same scale are averaged together to create the 8 scale scores.
  The eight health concepts are: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD. PhD., Principal Investigator — Professor
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sollie M, Thomsen JB, Sorensen JA. Autologous fat grafting seems to alleviate postherpetic neuralgia - a feasibility study investigating patient-reported levels of pain. J Plast Reconstr Aesthet Surg. 2021 Feb;74(2):350-356. doi: 10.1016/j.bjps.2020.08.038. Epub 2020 Aug 21. PMID 32917571
- [Derived] Sollie M, Sorensen JA. Treatment of chronic post-herpetic neuralgia with autologous fat grafts: a first-in-the-world case report. Br J Pain. 2019 Nov;13(4):239-243. doi: 10.1177/2049463718817570. Epub 2018 Nov 28. PMID 31656630